CLINICAL TRIAL: NCT01515397
Title: Efficacy and Safety of a Balanced Gelatine Solution in Combination With a Balanced Electrolyte Solution Versus a Standard Gelatine Solution in Combination With a Non-balanced Electrolyte Solution in Patients Scheduled for Abdominal Surgery
Brief Title: Comparison of Two Gelatine Solutions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC-G-H-0904
Record Dates: First submitted 2012-01-02; First posted 2012-01-24 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- balanced gelatine solution (Experimental): isotonic colloidal volume substitute
  Interventions: Drug: Gelofusine balanced
- non-balanced gelatine solution (Active Comparator): colloidal volume substitute
  Interventions: Drug: Gelofusine 4%

INTERVENTIONS:
Drug: Gelofusine balanced — Gelofusine balanced combined with Sterofundin ISO
  Arms: balanced gelatine solution
Drug: Gelofusine 4% — Gelofusine 4% combined with NaCl 0.9%
  Arms: non-balanced gelatine solution

SUMMARY:
The aim of volume replacement is to compensate a reduction in the intravascular volume e.g. during surgery and to counteract hypovolemia in order to maintain hemodynamics and vital functions. To achieve this, different plasma substitutes are available: Albumin, dextran, hydroxyethylstarches and gelatine. The aim of this study is to demonstrate that acid-base alterations during elective abdominal surgery can be reduced by the use of a new gelatine solution.

ELIGIBILITY:
Inclusion:

* Male or female patients >= 18 years of age and <= 90 years of age. Women of child bearing potential must test negative on standard pregnancy test.
* Patients scheduled to undergo elective abdominal surgery (e.g. Rectal resection, liver resection, open bowl resection, duodenopancreatectomy reconstitution).
* Scheduled intraoperative volume requirement of at least 15 ml / kg body weight (BROCA) gelatine solution
* Provision of voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent form approved by the Institutional Ethics Committee (IEC) prior to all evaluations.

Exclusion:

* Patients of ASA-class > III
* Known hypersensitivity to gelatine or to any of the constituents of the solution
* Patients treated with other colloid solutions and / or blood products 24 hours prior to surgery
* Patients on hemodialysis
* Patients suffering from decompensated renal function (i.e. serum creatinine > 3.0 mg/dl)
* Patients suffering from Hypervolemia Hyperhydration Severe blood coagulation disorders Hypernatremia (serum(Na+) > 150 mmol/L) Hyperchloremia (serum(Cl-) > 110 mmol/L)
* Estimated perioperative need for blood products of 3,5 ml / kg body weight (BROCA)
* Lactation period
* Simultaneous participation in another clinical trial
* Emergencies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
base excess [mmol/l] | Change from baseline at end of surgery, an expected average of 2 hours surgery
chloride [mmol/l] | Change from baseline at end of surgery, an expected average of 2 hours surgery

SECONDARY OUTCOMES:
arterial blood gase analyses | until 12 hours after surgery
coagulation status | until 12 hours after surgery
renal function | until 12 hours after surgery
adverse events | until 12 hours after surgery
hemodynamics (systolic and diastolic blood pressure) | until 12 hours after surgery
time on ventilation | until 12 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gernot Marx, Prof. Dr. med., Principal Investigator — Universitätsklinikum Aachen,Klinik für Operative Intensivmedizin
Locations (2):
- Germany (2):
  - Universitätsklinikum Aachen, Klinik für Anästhesiologie, Aachen
  - Klinik für Anästhesiologie, Intensivmedizin und Schmerztherapie, Universitätsklinikum Frankfurt/Main, Frankfurt am Main

REFERENCES:
- [Derived] Marx G, Meybohm P, Schuerholz T, Lotz G, Ledinko M, Schindler AW, Rossaint R, Zacharowski K. Impact of a new balanced gelatine on electrolytes and pH in the perioperative care. PLoS One. 2019 Apr 29;14(4):e0213057. doi: 10.1371/journal.pone.0213057. eCollection 2019. PMID 31034525